CLINICAL TRIAL: NCT06731751
Title: A Prospective, International Observational Study Assessing the Global Variation in Patient Characteristics, Management and Outcomes of Spontaneous Intracranial Haemorrhage.
Brief Title: The Planetary Outcomes After Intracranial Haemorrhage Study
Acronym: PLOT-ICH
Status: Not yet recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Sara Venturini, Miss, University of Cambridge
Other Study IDs: PLOTICH
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Intracerebral Haemorrhage; Subarachnoid Haemorrhage (SAH)
Keywords: brain haemorrhage; intracerebral haemorrhage; subarachnoid haemorrhage
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spontaneous Intracranial Haemorrhage Patients: Patients of any age with the presence of spontaneous intracranial haemorrhage (parenchymal, intraventricular and / or subarachnoid haemorrhage) on intracranial imaging (and absence of a history of trauma).
  Interventions: Other: Management of spontaneous intracranial haemorrhage

INTERVENTIONS:
Other: Management of spontaneous intracranial haemorrhage — Admission to hospital for spontaneous intracranial haemorrhage management. This includes admission for observation, conservative or interventional (surgical or endovascular) management to both ward-based and critical care settings.

SUMMARY:
Over twelve million strokes occur worldwide every year, and stroke is the second most common cause of death globally. Strokes happen because blood supply to the brain is damaged. This can be due to a blockage (ischaemic stroke) or a bleed (haemorrhagic stroke - or intracranial haemorrhage). Intracranial haemorrhage can be life-threatening and patients with this type of stroke can be very sick, requiring urgent medical care including medications, close monitoring, and sometimes surgery.

Strokes happen worldwide, but over 80% of stroke cases and associated death and disability occur in low- and middle- income countries (LMICs), where resources to manage them can be limited. However, the differences in how patients present, the hospital care they receive, and their overall outcomes when compared to high-income countries (HICs) patients are not fully understood. There are many stroke-related deaths occurring each year around the world, especially among those who have presented with an intracranial haemorrhage, and if survival rates are to be improved, high-quality data is needed to help us better understand where the improvements in care are required in different health settings.

Run and funded by the University of Cambridge, this study will collect data on all patients across all ages during a one-month period who undergo treatment for spontaneous intracranial haemorrhage, both medical and surgical. We will include patients from any hospital across the world that treats patients with this condition, collecting data from their admission to hospital until their discharge, death or up to 30 days from their presentation.

This is an observational study, so we are only observing patients care and management, not making any direct changes to their treatment. We will also be asking each centre to complete a written survey, to better understand some of the more complex areas which are important for the care of intracranial haemorrhage patients such as hospital resources available, and the potential barriers they face in accessing appropriate healthcare.

DETAILED DESCRIPTION:
Objectives Stroke is the second leading cause of death worldwide, with the greatest burden in LMICs. Haemorrhagic stroke or spontaneous intracranial haemorrhage (sICH), including intraparenchymal haemorrhage (IPH) and subarachnoid haemorrhage (SAH), has the greatest mortality and morbidity. Local management practices for haemorrhagic stroke vary greatly between geographical regions. This study aims to provide a comprehensive international overview of the patient characteristics, processes of care and short-term outcomes of patients being treated for sICH across high- and low-income settings.

Methods Study design: Prospective, international observational cohort study.

Setting: Any unit assessing patients with sICH is eligible to participate. Each participating unit will form a study team responsible for local approval processes, patient identification and data collection. Data will be collected online in anonymised form and will be analysed by the central study team according to a pre-determined statistical analysis plan.

Case definition:

Patients can be entered into the study if they meet the following criteria. • Patients of all ages with evidence of spontaneous intracranial haemorrhage (parenchymal, intraventricular and / or subarachnoid haemorrhage) on imaging (and absence of a history of trauma)

AND:

• Hospital admission for management of sICH All patients admitted to hospital meeting the above criteria during a given consecutive 30-day period during the study period will be included.

Results Data relating to the initial presentation, patient factors, management, and short-term outcomes of patients with sICH will be collected. The dataset includes patient demographics, details of the ictus, medical management, complications, timing and nature of surgical intervention (where applicable), post-intervention care and supporting management, and immediate post-operative complications. Primary outcome is 30-day mortality. Variation in processes of care and resources will be described. Where guidelines are available, outcomes will be assessed against guideline standards.

Conclusions This study aims to provide a global snapshot of the patient factors, management, processes of care and short-term outcomes of patients with spontaneous ICH and describe the global neurosurgical burden of haemorrhagic stroke. It will serve as a platform to facilitate future research and collaboration in global cerebrovascular surgery and stroke care.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with the presence of spontaneous intracranial haemorrhage (parenchymal, intraventricular and / or subarachnoid haemorrhage) on intracranial imaging (and absence of a history of trauma).

AND:

• Admission to hospital for sICH management. This includes admission for observation, conservative or interventional management to both ward-based and critical care settings.

Exclusion Criteria:

* Patients who have a clear history of trauma as the primary cause of the haemorrhage and therefore are diagnosed with traumatic intracranial haemorrhage.
* Patients with subdural or extradural haematomas but no clear history of trauma.
* Patients with intracranial haemorrhage occurring as a complication of a procedure or intervention (e.g. post-operative haematoma) or iatrogenic (e.g. after thrombolysis for ischaemic stroke).
* Patients who undergo elective (planned admission to hospital) or semi-elective (where a patient was initially admitted to hospital, then discharged from hospital and re-admitted for surgery) procedures.
* Patients re-admitted to hospital within 30 days of the initial admission with sICH (including those re-admitted for acute management of sICH-related complications).
* Patient presenting to the emergency department (ED) but discharged home from the ED immediately without a period of observation or admission to a ward.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult and paediatric patients meeting the case definition criteria and admitted to a participating institution with a sICH during the selected 30-day study period are eligible for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  30-day mortality or at discharge (whichever takes place first)

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
  Time in hospital, from admission to discharge
Complications | 30 days
  Peri-operative and disease specific complications (e.g. hydrocephalus, seizures, delayed cerebral ischaemia, return to operating theatre)
Modified Rankin Scale (mRS) | 30 days
  Modified Rankin Scale (mRS) as assessment of neurological function at discharge from hospital.
Glasgow Coma Scale | 30 days
  Glasgow Coma Scale (GCS) at discharge from hospital.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Venturini S, Clark D, Smith BG, Hobbs L, Bath MF, Mee H, Still M, Mediratta S, Soliman MA, Kohler K, Whiffin CJ, Katambo E, Korhonen TK, Tetri S, Bankole NDA, Rutabasibwa N, Bhebhe A, Munusamy T, Tirsit A, Park KB, Budohoski K, Wahjoepramono P, Tamborska A, Saylor D, Khan T, Khattak AF, Figaji A, Kolias AG, Bashford T, Joannides A, Martin M, Trivedi RA, Hutchinson PJ; PLOT-ICH Collaborative. Assessing the global variation in patient characteristics, management and short-term outcomes of spontaneous intracranial haemorrhage worldwide: a protocol for a global observational prospective multicentre study (the PLOT-ICH study). BMJ Open. 2025 Sep 2;15(9):e100361. doi: 10.1136/bmjopen-2025-100361. PMID 40897474